CLINICAL TRIAL: NCT02249780
Title: The Use of Indocyanine Green Fluorescence to Assses the Vascularisation of the Parathyroid Glands During Thyroid Surgery
Brief Title: Assessing Parathyroid Glands Vascularisation by ICG Fluoroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Geneva University, School of medicine (Unknown)
Responsible Party: Principal Investigator, JORDI VIDAL FORTUNY, Chef de clinique, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-160
Record Dates: First submitted 2014-09-15; First posted 2014-09-26 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2014-09

CONDITIONS: Parathyroid Function Low Adverse Event
Keywords: Parathyroid gland angiography; Parathyroid gland indocyanine green angiography; Parathyroid gland indocyanine green fluoroscopy
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- New treatment (Experimental): In patients with at least one well perfused parathyroid gland on ICG parathyroid angiography, no postoperative parathyroid dosage and supplementation will be done. Calcium and parathormone dosage will be done 10 days after surgery.
  Interventions: Procedure: No postoperative parathyroid dosage and supplementation; Procedure: ICG parathyroid angiography
- Standart treatment (Active Comparator): In those patients in whom at least on of the four parathyroid glands is well perused, postoperative parathyroid function test and parathyroid supplementation will be done. Calcium and parathormone dosage will be done at 24 hours and 10 days after surgery. Prophylactic supplementation of calcium and Vitamin D will be given.
  Interventions: Procedure: Postoperative parathyroid function test; Procedure: ICG parathyroid angiography; Drug: Parathyroid supplementation

INTERVENTIONS:
Procedure: Postoperative parathyroid function test — Calcium and parathormone dosage at 24 hours and ten day after surgery
  Arms: Standart treatment
Procedure: No postoperative parathyroid dosage and supplementation — The patients will be clinically followed for 24 hours after surgery and caclium and parathormone dosage will be done at ten days after surgery. No supplementation will be given.
  Other Names: Parathiroid function testing
  Arms: New treatment
Procedure: ICG parathyroid angiography — Injection of 3,5 mL of indocyanine green intravenously and perform angiography of parathyroid glands after thyroid removal.
  Other Names: Indoyanine green angiography; Indoyanine green fluoroscopy
Drug: Parathyroid supplementation — Supplementration with Calcimagon D3 Forte (1gr Calcium and 800 IU of 25-OH-vitamin D) from surgery day to up to 10 days afeter surgery.
  Other Names: Hypocalcemia post thyroidectomy treatment
  Arms: Standart treatment

SUMMARY:
Evaluate parathyroid gland perfusion during total thyroidectomy or thyroid totalisation surgery. Create an objective basis for the decision whether or not to transplant the parathyroid glands. Avoide postoperative serum calcium and parathyroid hormone dosages, and thus abstention of systematic supplementation with calcium and vitamin D in case of good perfusion.

DETAILED DESCRIPTION:
Parathyroid intraoperative indocyanine green (ICG) angiography is a new concept. To simplify the procedure the investigators have classified images into three categories: ICG 2: good blood supply (the gland has a white color); ICG 1: traumatic gland (the gland has a grayish color) and ICG 0: the gland is not vascularized (she has a black color). The investigators have applied the same criteria for visual values.

The investigators will randomize 138 patients with good ICG test values (at least one gland that is visually ≥1 and ICG 2): 69 will be subject to the usual postoperative care in the investigators service: 24 hours monitoring with dosage of calcium and PTH in the morning on postoperative day 1 and routine supplementation with Calcimagon D3 Forte (1g Calcium and 800 IU of 25-OH-vitamin D) BD by mouth until postoperative follow-up appointment, which takes place between day 10 and 15. Depending on the results of blood tests patients will also be given Rocaltrol substitution (1, 25-OH-Vitamin D) 0.5mcg BD. The remaining patients will be monitored 24 hours in hospital looking for clinical signs and symptoms of hypocalcemia but without any blood dosage or systematic supplementation. If signs and / or symptoms of hypocalcemia develop (tingling, muscle spasms, Chvostek sign), a blood test will be performed and patients will be substituted by the usual protocol. All patients will be reviewed at 10 - 15 days of the intervention with the relevant balance sheet.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing total thyroidectomy or a totalisation thyroid procedure.
* Patients capable of understanding and able to understand the study.
* Values visually 2 and ICG 2

Exclusion Criteria:

* Parathyroid disease or prior parathyroidectomy
* Lack of informed consent
* Altered mental status of the patient.
* ICG values <2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Postoperative parathyroid function | 10 days after surgery
  All patients will be reviewed at 10-15 days after surgery and blood tests will be done. Investigators will check the number of patients with serum calcium and parathyroid hormone in normal ranges at ten days after surgery in both arms of the study. Low parathyroid function will be diagnosed when corrected calcium < 2mmol/l, and PTH < 1.1 pmol/l.

SECONDARY OUTCOMES:
Calcium and parathormone dosage after surgery | 10 days after surgery
  Number of patients with good calcium and parathormone values at 10 days after surgery without calcium and vitamin D supplementation in the selected group.

OTHER OUTCOMES:
Economic impact | From surgery day to 10 days after surgery
  Compare the costs of both procedures: standard procedure and new treatment and then evaluate the economic impact of this preventig mesure, and the possibility to undergo ambulatory surgery

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Triponez, Professor, Study Director — University Hospital, Geneva; Wolfram Karenovics, SPR, Principal Investigator — University Hospital, Geneva; Frédéric Ris, Consultant, Principal Investigator — University Hospital, Geneva; Valentina Belfontali, Resident, Principal Investigator — University Hospital, Geneva; Jordi Vidal Fortuny, SPR, Study Chair — University Hospital, Geneva
Locations (1):
- University Hospitals Geneva, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Vidal Fortuny J, Sadowski SM, Belfontali V, Guigard S, Poncet A, Ris F, Karenovics W, Triponez F. Randomized clinical trial of intraoperative parathyroid gland angiography with indocyanine green fluorescence predicting parathyroid function after thyroid surgery. Br J Surg. 2018 Mar;105(4):350-357. doi: 10.1002/bjs.10783. Epub 2018 Feb 6. PMID 29405252